CLINICAL TRIAL: NCT01691820
Title: A Study in Adolescent Females to Explore Cytomegalovirus Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 115639
Record Dates: First submitted 2012-09-13; First posted 2012-09-25 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Infections, Cytomegalovirus
Keywords: Adolescent females; Cytomegalovirus (CMV)
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Blood Specimen Collection; Urine Specimen Collection

ARMS (3):
- Group S+ (Experimental): Cytomegalovirus (CMV) seropositive subjects aged between 10-17 years at enrollment in the study.
  Interventions: Procedure: Blood collection; Procedure: Urine collection; Procedure: Saliva collection
- Group S- (Experimental): Cytomegalovirus (CMV) seronegative subjects aged between 10-17 years at enrollment in the study.
  Interventions: Procedure: Blood collection; Procedure: Urine collection; Procedure: Saliva collection
- Missing serostatus Group (Experimental): Subjects with no confirmed serostatus, aged between 10-17 years at enrollment in the study.
  Interventions: Procedure: Blood collection; Procedure: Urine collection; Procedure: Saliva collection

INTERVENTIONS:
Procedure: Blood collection — Samples collected at Months 0, 4, 8, 12, 16, 20, 24, 28, 32, and 36.
Procedure: Urine collection — Samples collected at Months 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 34, and 36.
Procedure: Saliva collection — Samples collected at Months 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 34, and 36.

SUMMARY:
The purpose of this study is to estimate the incidence of Cytomegalovirus (CMV) secondary infections (re-infections/re-activations) and the incidence of CMV primary infections in adolescent females.

ELIGIBILITY:
Inclusion Criteria:

* A female adolescent between, and including 10 and 17 years at the time of enrolment regardless of pregnancy status and contraception method used or not used.
* Subjects who the investigator believes that the subject and/or the subject's parent(s)/Legally Acceptable Representative(s) (LAR[s]) can and will comply with the requirements of the protocol.
* Written informed assent and/or consent obtained from the subject and/or the parent(s)/LAR(s) of the subject.
* Subject is likely to remain in the area and/or return for required study Site Visits and complete Sample Collection Visits.

Exclusion Criteria:

* Child in care.
* Use or planned use of any investigational or non-registered antiviral drug or vaccine during the study period.
* Known medical history of any recurrent clinical herpes episodes requiring episodic or chronic suppressive treatment with oral or parenteral antiviral treatment such as acyclovir, famciclovir, valacyclovir or any other anti-herpes virus anti-viral during the year preceding enrolment. Topical anti-viral are allowed.
* Subjects with history of previous vaccination against CMV.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to Visit 1 or planned administration during the study. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products within 3 months prior to Visit 1 or planned administration during the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including HIV-infection, based on medical history and physical examination (no laboratory testing required).
* Any major congenital defects, serious chronic illness or organ transplantation.

Ages: 10 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 369 (Actual)
Dates: Start 2012-10-05 (Actual); Primary Completion 2017-04-08 (Actual); Study Completion 2017-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (2):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Stevensville, Michigan
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Oulu
- GSK Investigational Site, Jojutla, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paris R, Apter D, Boppana S, D'Aloia M, De Schrevel N, Delroisse JM, Grassano L, Guignard A, Panackal AA, Roman F, Yu J, Yunes EM, Dieussaert I. Incidence of Cytomegalovirus Primary and Secondary Infection in Adolescent Girls: Results From a Prospective Study. J Infect Dis. 2023 Nov 28;228(11):1491-1495. doi: 10.1093/infdis/jiad182. PMID 37340664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolment was terminated once approximately 240 seropositive subjects were included in the trial, to obtain approximately 200 evaluable seropositive subjects. The number of seronegative subjects enrolled depended on the seroprevalence of the participating countries.
Pre-assignment Details: Of the 369 enrolled subjects, 363 were female subjects and 6 were newborns of some subjects. Consent was signed for the newborns to allow testing for CMV disease. The objectives assessed the CMV infections in the adolescent females with a known serostatus (N=362); no demographics, outcome measures, or adverse events were assessed in newborns.
Period: Overall Study
Arm/Group | Group S+ | Group S-
Started | 210 | 152
Completed | 184 | 115
Not Completed | 26 | 37
Not completed — Consent withdrawal (not due to an AE) | 9 | 15
Not completed — Migrated/moved from study area | 7 | 4
Not completed — Lost to Follow-up | 6 | 17
Not completed — Other (unspecified) | 4 | 1

BASELINE CHARACTERISTICS:
Population: The primary and secondary objectives of this study have assessed the incidence of CMV infections in adolescent females only, hence no demographic data was collected for the 6 newborns.
Groups:
- Group S+: CMV seropositive subjects, aged 10-17 years at enrollment in the study.
- Group S-: CMV seronegative subjects, aged 10-17 years at enrollment in the study.
- Total: Total of all reporting groups
Arm/Group | Group S+ | Group S- | Total
Number analyzed (Participants) | 210 | 152 | 362
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.5 (2.1) | 13.4 (2.2) | 13.5 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 152 | 362
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 8 | 8 | 16
  Asian - South East Asian Heritage | 1 | 0 | 1
  White - Arabic / North African Heritage | 0 | 1 | 1
  White - Caucasian / European Heritage | 64 | 93 | 157
  Other | 137 | 50 | 187

OUTCOME MEASURES:

1. Primary Outcome: Number of CMV Seropositive Subjects With Appearance or Increase of Anti-CMV Tegument Protein IgG Antibodies in Serum.
Description: This outcome was part of the assessment of occurrence of CMV secondary infections determined in all seropositive subjects. Two-fold and above increases" category = subjects that had two-fold and above increases of anti-CMV Immunoglobulin G (IgG) concentration. "Four-fold and above increases" = subjects that had four-fold and above increases of anti-CMV IgG concentration. The cut-off of the assay = 1.136 ELISA unit (EU)/mL. A seropositive subject is a subject for whom anti-CMV IgG antibodies were detected in serum sample collected at Month 0. CMV secondary infections are defined as either a viral reactivation or a re-infection with a new strain of CMV.
Time Frame: At Month 4
Population: This analysis was performed on CMV seropositive subjects with available results at Month 4 from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Count of Participants; unit: Participants
Groups:
- Group S+: CMV seropositive subjects aged between 10-17 years at enrollment in the study.
Arm/Group | Group S+
Number analyzed (Participants) | 202
Participants
  anti-Teg IgG - Two-fold and above increases | 5
  anti-Teg IgG -Four-fold and above increases | 2

2. Primary Outcome: Number of CMV Seropositive Subjects With Appearance or Increase of Anti-CMV Tegument Protein IgG Antibodies in Serum.
Description: This outcome was part of the assessment of occurrence of CMV secondary infections determined in all seropositive subjects. Two-fold and above increases" category = subjects that had two-fold and above increases of anti-CMV IgG concentration. "Four-fold and above increases" = subjects that had four-fold and above increases of anti-CMV IgG concentration. The cut-off of the assay = 1.136 ELISA unit (EU)/mL. A seropositive subject is a subject for whom anti-CMV IgG antibodies were detected in serum sample collected at Month 0. CMV secondary infections are defined as either a viral reactivation or a re-infection with a new strain of CMV.
Time Frame: At Month 8
Population: This analysis was performed on CMV seropositive subjects with available results at Month 8 from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Count of Participants; unit: Participants
Groups:
- Group S+: CMV seropositive subjects aged between 10-17 years at enrolment in the study.
Arm/Group | Group S+
Number analyzed (Participants) | 197
Participants
  Two-fold and above increases | 5
  Four-fold and above increases | 1

3. Primary Outcome: Number of CMV Seropositive Subjects With Appearance or Increase of Anti-CMV Tegument Protein IgG Antibodies in Serum.
Description: as for outcome 2
Time Frame: At Month 12
Population: This analysis was performed on CMV seropositive subjects with available results at Month 12 from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Group S+
Number analyzed (Participants) | 198
Participants
  Two-fold and above increases | 6
  Four-fold and above increases | 3

4. Primary Outcome: Number of CMV Seropositive Subjects With Appearance or Increase of Anti-CMV Tegument Protein IgG Antibodies in Serum.
Description: as for outcome 2
Time Frame: At Month 16
Population: This analysis was performed on CMV seropositive subjects with available results at Month 16 from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Group S+
Number analyzed (Participants) | 196
Participants
  Two-fold and above increases | 1
  Four-fold and above increases | 0

5. Primary Outcome: Number of CMV Seropositive Subjects With Appearance or Increase of Anti-CMV Tegument Protein IgG Antibodies in Serum.
Description: as for outcome 2
Time Frame: At Month 20
Population: This analysis was performed on CMV seropositive subjects with available results at Month 20 from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Group S+
Number analyzed (Participants) | 191
Participants
  Two-fold and above increases | 5
  Four-fold and above increases | 2

6. Primary Outcome: Number of CMV Seropositive Subjects With Appearance or Increase of Anti-CMV Tegument Protein IgG Antibodies in Serum.
Description: as for outcome 2
Time Frame: At Month 24
Population: This analysis was performed on CMV seropositive subjects with available results at Month 24 from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Group S+
Number analyzed (Participants) | 189
Participants
  Two-fold and above increases | 6
  Four-fold and above increases | 2

7. Primary Outcome: Number of CMV Seropositive Subjects With Appearance or Increase of Anti-CMV Tegument Protein IgG Antibodies in Serum.
Description: as for outcome 2
Time Frame: At Month 28
Population: This analysis was performed on CMV seropositive subjects with available results at Month 28 from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Group S+
Number analyzed (Participants) | 188
Participants
  Two-fold and above increases | 5
  Four-fold and above increases | 1

8. Primary Outcome: Number of CMV Seropositive Subjects With Appearance or Increase of Anti-CMV Tegument Protein IgG Antibodies in Serum.
Description: as for outcome 2
Time Frame: At Month 32
Population: This analysis was performed on CMV seropositive subjects with available results at Month 32 from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Group S+
Number analyzed (Participants) | 184
Participants
  Two-fold and above increases | 1
  Four-fold and above increases | 1

9. Primary Outcome: Number of CMV Seropositive Subjects With Appearance or Increase of Anti-CMV Tegument Protein IgG Antibodies in Serum.
Description: as for outcome 2
Time Frame: At Month 36
Population: This analysis was performed on CMV seropositive subjects with available results at Month 36 from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Group S+
Number analyzed (Participants) | 180
Participants
  Two-fold and above increases | 3
  Four-fold and above increases | 0

10. Primary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentration in Serum (ELISA).
Description: This outcome was part of the assessment of occurrence of CMV secondary infections determined in all seropositive subjects. A seropositive subject is a subject for whom anti-CMV IgG antibodies were detected in serum sample collected at Month 0. CMV secondary infections are defined as either a viral reactivation or a re-infection with a new strain of CMV. Antibody concentrations were tabulated as geometric mean concentrations (GMC) and expressed as ELISA units (EU)/mL. The cut-off of the assay = 1.136 EU/mL.
Time Frame: At Month 0
Population: This analysis was performed on CMV seropositive subjects with available results at Month 0 from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group S+
Number analyzed (Participants) | 206
EU/mL | 5.4 [4.9 to 6.1]

11. Primary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentration in Serum (ELISA).
Description: This outcome was part of the assessment of occurrence of CMV secondary infections determined in all seropositive subjects. A seropositive subject is a subject for whom anti-CMV IgG antibodies were detected in serum sample collected at Month 0. CMV secondary infections are defined as either a viral reactivation or a re-infection with a new strain of CMV. Antibody concentrations were tabulated as geometric mean concentrations (GMC) and expressed as ELISA units (EU)/mL. The cut-off of the assay = 1.136 EU/mL. GMC was calculated on subjects meeting a two-fold increase or above (i.e.: subjects that had two-fold and above increases [including four-fold] of CMV anti-tegument IgG compared with previous time point).
Time Frame: At Month 4
Population: This analysis was performed on CMV seropositive subjects with available results and meeting the two-fold increase or above, at Month 4, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Groups:
- Group S+: CMV seropositive subjects, aged between 10-17 years at enrollment in the study.
Arm/Group | Group S+
Number analyzed (Participants) | 5
EU/mL | 32.2 [14.4 to 72.0]

12. Primary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentration in Serum (ELISA).
Description: as for outcome 11
Time Frame: At Month 8
Population: This analysis was performed on CMV seropositive subjects with available results and meeting the two-fold increase or above, at Month 8, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group S+
Number analyzed (Participants) | 5
EU/mL | 10.3 [2.8 to 38.0]

13. Primary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentration in Serum (ELISA).
Description: as for outcome 11
Time Frame: At Month 12
Population: This analysis was performed on CMV seropositive subjects with available results and meeting the two-fold increase or above, at Month 12, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group S+
Number analyzed (Participants) | 6
EU/mL | 9.8 [2.7 to 34.9]

14. Primary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentration in Serum (ELISA).
Description: as for outcome 11
Time Frame: At Month 16
Population: This analysis was performed on CMV seropositive subjects with available results and meeting the two-fold increase or above, at Month 16, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group S+
Number analyzed (Participants) | 1
EU/mL | 26.5 [NA to NA] — No Upper or Lower limits could be computed since there was only 1 subject who met the criterion.

15. Primary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentration in Serum (ELISA).
Description: as for outcome 11
Time Frame: At Month 20
Population: This analysis was performed on CMV seropositive subjects with available results and meeting the two-fold increase or above, at Month 20, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group S+
Number analyzed (Participants) | 5
EU/mL | 10.1 [3.7 to 27.7]

16. Primary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentration in Serum (ELISA).
Description: as for outcome 11
Time Frame: At Month 24
Population: This analysis was performed on CMV seropositive subjects with available results and meeting the two-fold increase or above, at Month 24, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group S+
Number analyzed (Participants) | 6
EU/mL | 9.3 [5.4 to 16.0]

17. Primary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentration in Serum (ELISA).
Description: as for outcome 11
Time Frame: At Month 28
Population: This analysis was performed on CMV seropositive subjects with available results and meeting the two-fold increase or above, at Month 28, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group S+
Number analyzed (Participants) | 5
EU/mL | 8.3 [2.4 to 28.9]

18. Primary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentration in Serum (ELISA).
Description: as for outcome 11
Time Frame: At Month 32
Population: This analysis was performed on CMV seropositive subjects with available results and meeting the two-fold increase or above, at Month 32, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group S+
Number analyzed (Participants) | 1
EU/mL | 14.4 [NA to NA] — No Upper or Lower limits could be computed since there was only 1 subject who met the criterion.

19. Primary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentration in Serum (ELISA).
Description: as for outcome 11
Time Frame: At Month 36
Population: This analysis was performed on CMV seropositive subjects with available results and meeting the two-fold increase or above, at Month 36, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group S+
Number analyzed (Participants) | 3
EU/mL | 6.9 [2.0 to 23.8]

20. Primary Outcome: Geometric Mean CMVpp65 Antibody Concentration in Subjects Based on Number of CMV Deoxyribonucleic Acid (DNA) Copies (pp65 Gene) in Urine
Description: This outcome was part of the assessment of occurrence of CMV secondary infections determined in all seropositive subjects. The concentration of DNA copies was assessed by quantitative Polymerase Chain Reaction (qPCR), for CMV seropositive subjects with appearance of CMV DNA (>0 copies/mL) and DNA copies=0 in prior urine sample (category="> 0 Copies/mL") and for CMV seropositive subjects with increase of CMV DNA (≥6720 copies/mL) and 0<DNA copies <LLOQ (6720 copies/mL) in prior urine sample (category name= "≥6720 copies/mL").
Time Frame: At Month 4
Population: This analysis was performed on the seropositive subjects with DNA copies data in prior urine sample and with CMV DNA copies above the specified cut-off, at Month 4, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: DNA copies/mL
Arm/Group | Group S+
Number analyzed (Participants) | 8
DNA copies/mL
  > 0 Copies/mL: number analyzed (Participants) | 7
  > 0 Copies/mL | 754.1 [144.6 to 3932.9]
  ≥ 6720 Copies/mL: number analyzed (Participants) | 1
  ≥ 6720 Copies/mL | 8310.0 [NA to NA] — No Upper or Lower limits could be computed since there was only 1 subject in this category.

21. Primary Outcome: Geometric Mean CMVpp65 Antibody Concentration in Subjects Based on Number of CMV DNA Copies (pp65 Gene) in Urine
Description: This outcome was part of the assessment of occurrence of CMV secondary infections determined in all seropositive subjects. The concentration of DNA copies was assessed by quantitative Polymerase Chain Reaction (qPCR),for CMV seropositive subjects with appearance of CMV DNA (>0 copies/mL) and DNA copies=0 in prior urine sample (category="> 0 Copies/mL") and for CMV seropositive subjects with increase of CMV DNA (≥6720 copies/mL) and 0<DNA copies <LLOQ (6720 copies/mL) in prior urine sample (category name= "≥6720 copies/mL").
Time Frame: At Month 8
Population: This analysis was performed on the seropositive subjects with DNA copies data in prior urine sample and with CMV DNA copies above the specified cut-off, at Month 8, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: DNA copies/mL
Groups:
- Group S+: CCMV seropositive subjects aged between 10-17 years at enrollment in the study.
Arm/Group | Group S+
Number analyzed (Participants) | 11
DNA copies/mL
  > 0 Copies/mL: number analyzed (Participants) | 10
  > 0 Copies/mL | 361.5 [166.9 to 783.3]
  ≥ 6720 Copies/mL: number analyzed (Participants) | 1
  ≥ 6720 Copies/mL | 15386.0 [NA to NA] — No Upper or Lower limits could be computed since there was only 1 subject in this category.

22. Primary Outcome: Geometric Mean CMVpp65 Antibody Concentration in Subjects Based on Number of CMV DNA Copies (pp65 Gene) in Urine
Description: This outcome was part of the assessment of occurrence of CMV secondary infections determined in all seropositive subjects. The concentration of DNA copies was assessed by quantitative Polymerase Chain Reaction (qPCR),for CMV seropositive subjects with appearance of CMV DNA (>0 copies/mL) and DNA copies=0 in prior urine sample (category="> 0 Copies/mL").
Time Frame: At Month 12
Population: This analysis was performed on the seropositive subjects with DNA copies data in prior urine sample and with CMV DNA copies above the specified cut-off, at Month 12, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures
Measure: Geometric Mean (95% Confidence Interval); unit: DNA copies/mL
Groups:
- Group S+: CMV seropositive, adolescent females aged between 10 and 17 years at enrollment in the study.
Arm/Group | Group S+
Number analyzed (Participants) | 10
DNA copies/mL | 647.4 [213.1 to 1966.6]

23. Primary Outcome: Geometric Mean CMVpp65 Antibody Concentration in Subjects Based on Number of CMV DNA Copies (pp65 Gene) in Urine
Description: as for outcome 22
Time Frame: At Month 16
Population: This analysis was performed on the seropositive subjects with DNA copies data in prior urine sample and with CMV DNA copies above the specified cut-off, at Month 16, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures
Measure: Geometric Mean (95% Confidence Interval); unit: DNA copies/mL
Arm/Group | Group S+
Number analyzed (Participants) | 9
DNA copies/mL | 348.7 [129.8 to 936.9]

24. Primary Outcome: Geometric Mean CMVpp65 Antibody Concentration in Subjects Based on Number of CMV DNA Copies (pp65 Gene) in Urine
Description: as for outcome 22
Time Frame: At Month 20
Population: This analysis was performed on the seropositive subjects with DNA copies data in prior urine sample and with CMV DNA copies above the specified cut-off, at Month 20, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures
Measure: Geometric Mean (95% Confidence Interval); unit: DNA copies/mL
Arm/Group | Group S+
Number analyzed (Participants) | 3
DNA copies/mL | 199.4 [97.5 to 408.0]

25. Primary Outcome: Geometric Mean CMVpp65 Antibody Concentration in Subjects Based on Number of CMV DNA Copies (pp65 Gene) in Urine
Description: as for outcome 22
Time Frame: At Month 24
Population: This analysis was performed on the seropositive subjects with DNA copies data in prior urine sample and with CMV DNA copies above the specified cut-off, at Month 24,from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures
Measure: Geometric Mean (95% Confidence Interval); unit: DNA copies/mL
Arm/Group | Group S+
Number analyzed (Participants) | 8
DNA copies/mL | 322.1 [112.8 to 919.4]

26. Primary Outcome: Geometric Mean CMVpp65 Antibody Concentration in Subjects Based on Number of CMV DNA Copies (pp65 Gene) in Urine
Description: as for outcome 21
Time Frame: At Month 28
Population: This analysis was performed on the seropositive subjects with DNA copies data in prior urine sample and with CMV DNA copies above the specified cut-off, at Month 28,from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures
Measure: Geometric Mean (95% Confidence Interval); unit: DNA copies/mL
Arm/Group | Group S+
Number analyzed (Participants) | 7
DNA copies/mL
  > 0 Copies/mL: number analyzed (Participants) | 6
  > 0 Copies/mL | 421.9 [71.3 to 2497.2]
  ≥ 6720 Copies/mL: number analyzed (Participants) | 1
  ≥ 6720 Copies/mL | 7369.0 [NA to NA] — No Upper or Lower limits could be computed since there was only 1 subject in this category.

27. Primary Outcome: Geometric Mean CMVpp65 Antibody Concentration in Subjects Based on Number of CMV DNA Copies (pp65 Gene) in Urine
Description: as for outcome 22
Time Frame: At Month 32
Population: This analysis was performed on the seropositive subjects with DNA copies data in prior urine sample and with CMV DNA copies above the specified cut-off, at Month 32, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures
Measure: Geometric Mean (95% Confidence Interval); unit: DNA copies/mL
Arm/Group | Group S+
Number analyzed (Participants) | 3
DNA copies/mL | 186.1 [15.0 to 2308.8]

28. Primary Outcome: Geometric Mean CMVpp65 Antibody Concentration in Subjects Based on Number of CMV DNA Copies (pp65 Gene) in Urine
Description: as for outcome 22
Time Frame: At Month 36
Population: This analysis was performed on the seropositive subjects with DNA copies data in prior urine sample and with CMV DNA copies above the specified cut-off, at Month 36, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures
Measure: Geometric Mean (95% Confidence Interval); unit: DNA copies/mL
Arm/Group | Group S+
Number analyzed (Participants) | 7
DNA copies/mL | 915.3 [123.0 to 6808.7]

29. Secondary Outcome: Number of CMV Seronegative Subjects With Appearance of Anti-CMV Tegument Protein IgG Antibodies in Serum.
Description: This outcome was part of the assessment of occurrence of CMV primary infections determined in all seronegative subjects, on samples collected during the 4-month site visits until study conclusion. A seronegative subject is a subject for whom anti-CMV IgG antibodies were not detected in serum sample collected at Month 0. CMV primary infection is defined as the first infection with CMV in subjects who were seronegative at enrollment.
Time Frame: From study Month 0 to Month 36
Population: This analysis was performed on the seronegative subjects with available results at the specified timepoints, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Count of Participants; unit: Participants
Groups:
- Group S-: CMV seronegative subjects, aged between 10-17 years at enrollment in the study.
Arm/Group | Group S-
Number analyzed (Participants) | 152
Participants
  Month 0 | 0
  Month 4: number analyzed (Participants) | 143
  Month 4 | 5
  Month 8: number analyzed (Participants) | 142
  Month 8 | 5
  Month 12: number analyzed (Participants) | 142
  Month 12 | 4
  Month 16: number analyzed (Participants) | 137
  Month 16 | 6
  Month 20: number analyzed (Participants) | 129
  Month 20 | 8
  Month 24: number analyzed (Participants) | 134
  Month 24 | 12
  Month 28: number analyzed (Participants) | 126
  Month 28 | 8
  Month 32: number analyzed (Participants) | 122
  Month 32 | 9
  Month 36: number analyzed (Participants) | 113
  Month 36 | 12

30. Secondary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentration of Seronegative Subjects
Description: This outcome is part of the assessment of occurrence of CMV primary infections determined in all seronegative subjects, on samples collected during the 4-month site visits until study conclusion. A seronegatve subject is a subject for whom anti-CMV IgG antibodies were not detected in serum sample collected at Month 0. CMV primary infection is defined as the first infection with CMV in subjects who were seronegative at enrollment. Antibody concentrations were tabulated as geometric mean concentrations (GMC) and expressed as ELISA units (EU)/mL. The cut-off of the assay = 1.136 EU/mL.
Time Frame: From study Month 0 to Month 36
Population: This analysis was performed on the seronegative subjects with available results at Month 0, or on the seronegative subjects with antibody concentration above 1.136 U/mL for the other time points, from the According-to-Protocol cohort, which included all subjects who met all inclusion criteria and no exclusion criteria for the study, who did not have any elimination criteria during the study and who complied with the study procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group S-
Number analyzed (Participants) | 152
EU/mL
  Month 0 | 0.4 [0.3 to 0.4]
  Month 4: number analyzed (Participants) | 5
  Month 4 | 2.4 [0.8 to 7.2]
  Month 8: number analyzed (Participants) | 5
  Month 8 | 2.6 [0.8 to 9.0]
  Month 12: number analyzed (Participants) | 4
  Month 12 | 1.8 [0.5 to 6.7]
  Month 16: number analyzed (Participants) | 6
  Month 16 | 3.5 [1.2 to 9.8]
  Month 20: number analyzed (Participants) | 8
  Month 20 | 4.5 [2.2 to 9.3]
  Month 24: number analyzed (Participants) | 12
  Month 24 | 2.7 [1.5 to 5.0]
  Month 28: number analyzed (Participants) | 8
  Month 28 | 3.5 [1.4 to 8.4]
  Month 32: number analyzed (Participants) | 9
  Month 32 | 3.4 [1.7 to 7.1]
  Month 36: number analyzed (Participants) | 12
  Month 36 | 4.5 [2.1 to 9.6]

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected throughout the entire study, from Month 0 up to Month 36.
Description: There were no Other (Not Including Serious) Adverse Events collected in this study, as there were no vaccines administered.
Groups:
- Group S+: CMV seropositive subjects aged 10-17 years at enrollment in the study.
- Group S-: CMV seronegative subjects aged 10-17 years at enrollment in the study.
Arm/Group | Group S+ | Group S-
All-Cause Mortality (participants affected / at risk) | 0/210 | 0/152
Serious Adverse Events (participants affected / at risk) | 0/210 | 0/152
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-02-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT01691820/Prot_001.pdf
  • Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT01691820/SAP_000.pdf